CLINICAL TRIAL: NCT05316012
Title: The Integration of Sensor Technology Into Incontinence Materials: a Single-group Pretest-posttest Study in a Nursing Home Environment
Acronym: Smart Diapers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BC-09902
Record Dates: First submitted 2022-02-22; First posted 2022-04-07 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Incontinence
Keywords: incontinence; sensor technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Residents (Experimental): 5 residents - fase 1 Intervention device: smart diaper (diaper, sensor and strips, without alerting system).
  15 residents -fase 2, of which 5 residents of study phase 1 Intervention device: smart diaper (diaper, sensor and strips, with alerting system)
  Interventions: Device: Smart diapers

INTERVENTIONS:
Device: Smart diapers — Residents receive standard continence care while using the smart diaper (without the alerting system) - fase 1
  Diapers are changed as usual, e.g., after morning care, visual soiling, unpleasant odor, saturation, leakage.
  Residents receive continence care while using the smart diaper with the alerting system - fase 2

SUMMARY:
The smart diaper aims to (1) detect humidity, (2) be capable of sending real-time indication of the saturation to the healthcare workers when urine loss occurs and (3) generate alerts when the diaper requires changing. Potential benefits of the smart diaper compared to incontinence management products without sensor technology include: workload reduction, increased comfort for residents and staff, more person-centred care, increased quality of care, less skin damage and economic (e.g. less costs due to less excessive diaper changes), and/or environmental (e.g. less waste) gains.

ELIGIBILITY:
Inclusion Criteria:

* Resident of nursing home
* Urinary incontinence or double incontinence (Katz score incontinence ≥ 3) by day and night. (Score assessed in one week interval before start study period 1 and 2 "D1")
* Wearing adult diapers as incontinence material, size M.
* Unable to change diaper independently when saturated or leaking (Katz score toileting ≥ 3). (Score assessed in one week interval before start study period 1 and 2 "D1")
* Written informed consent from resident or resident's legal representative.
* Dutch speaking

Exclusion Criteria:

* Residents who are receiving end-of-life care
* Residents with a Mini-Mental State Examination (MMSE)-score of < 24
* Residents with a dominant belly sleeping position

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-11-27 (Actual)

PRIMARY OUTCOMES:
Mean percentage saturation | 10 days
  The difference between the percentage saturation determined by the smart diaper and the percentage saturation based on the data registered in the frequency volume urine charts (FVUCs) (during each study period* for each diaper change)
The % of correct warnings | 10 days
  = warning on saturation of the incontinence material) generated by the sensor.
  a. Each warning generated by the sensor will be assessed by the nurse (correct/incorrect warning)
Frequency of skin irritations | 10 days
  3. The frequency of skin irritations related to incontinence (Incontinence-Associated Dermatitis or IAD) in the gluteal/sacral area (assessed daily during each study period*).

CONTACTS AND LOCATIONS:
Locations (1):
- WZC Heilig Hart vzw, Oudenaarde, Belgium

IPD SHARING:
Plan to Share IPD: No